CLINICAL TRIAL: NCT01391442
Title: Family Heritability, Investigating Gene-gene and Gene-environment Interactions in the Field of Cardiovascular Diseases - 4th VISIT (at 17 Years) of the STANISLAS COHORT
Brief Title: - 4th Visit at 17 Years of Cohort STANISLAS - Stanislas Ancillary Study ESCIF
Acronym: STANISLASV4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pr. Nicolas GIRERD (Other)
Responsible Party: Sponsor-Investigator, Pr. Nicolas GIRERD, Clinical Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010-A01469-30
Record Dates: First submitted 2011-05-12; First posted 2011-07-12 (Estimated); Last update posted 2024-03-28 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases
Keywords: follow up of troop,; MRI, Echocardiography, Functional indices
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Blood Specimen Collection; Biological Oxygen Demand Analysis; Heart Disease Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- family (Other): each family, composed of 4 characters at least, is studied
  Interventions: Biological: blood and urine samples; Genetic: blood sample; Other: cardiovascular assessment; Other: Stanislas ancillary study : MRI examination with GRICS technique

INTERVENTIONS:
Biological: blood and urine samples — 58 ml of blood 120 ml of urine
  Other Names: biological analyses; biological collection
Genetic: blood sample — 11 ml of blood
  Other Names: ADN and ARN collection
Other: cardiovascular assessment — echography, echodoppler, measure of blood pressure...
  Other Names: cardiovascular risk factors
Other: Stanislas ancillary study : MRI examination with GRICS technique

SUMMARY:
The Stanislas Cohort is a monocentric familial longitudinal cohort comprised of 1006 families (4295 subjects) from the Nancy region recruited in 1993-1995 at the Centre for Preventive Medicine (Centre de Médecine Préventive, CMP), Vandoeuvre lès Nancy for a 5-year periodic health examination, under the auspices of the Caisse Nationale d'Assurance Maladie (CNAM).

This cohort was established with the primary objective of investigating gene-gene and gene-environment interactions in the field of cardiovascular diseases, based on the study of inter-individual variability and familial segregation analysis of biological and morphological intermediate phenotypes of cardiovascular risk. The longitudinal nature of this study should enable to take into account the evolution of intermediate phenotypes related to genetic factors throughout the follow-up period. The families, consisting of two parents and at least two biological children, were deemed healthy, free of declared acute and/or chronic illness, in order to assess the effect of genetics on the variability of intermediate phenotypes studied under physiological conditions (without the influence, in the absence) of pathology.

The Stanislas Cohort is, both nationally and internationally, the only longitudinal familial cohort of supposedly healthy subjects on such a large scale.

Brief summary of ancillary study "Cardiac Functional Indices Comparison Between MRI and Echocardiography" : the ESCIF study is an ancillary study of the Stanislas cohort aiming at comparing in a cohort of supposedly healthy subjects different cardiac functional indices between two different modalities : Echocardiography and MRI. Indeed, new cardiac functional indices have been recently developed in the scope of echocardiography and would be very useful in MRI. In echography they are computed either from tissue Doppler imaging or from a specific image analysis called speckle tracking. These two techniques are accessible in MRI with the Generalized Reconstruction by Inversion of Coupled Systems (GRICS) technology which provides a motion model from which strains and strain rates may be derived and which allow longer acquisition without the constraint of breath holding (mandatory to reach high temporal resolution).

DETAILED DESCRIPTION:
MAIN STUDY Follow-up visit No. 4 is currently being scheduled, and is planned between 2011 and 2016.

Objectives:

* Conduct a fourth visit, in 2011-2016, enabling a follow-up at 17 years of the cohort population.
* Enrich the sample collection with new biobanks and clinical phenotyping of the cohort by conducting selected specific investigations and supported by specific scientific hypotheses and protocols
* Evaluate the long-term (follow-up, monitoring) of clinical, biological, morphological data by analyzing:

  * The influence of aging (average age of parents in 1993: 45 years and in 2010-2012: 62 years).
  * The incidence and changes in prevalence of cardiovascular risk factors comprising the metabolic syndrome (MS), and their familial segregation, since as early as the second visit, in some one hundred families, at least one family member presented a MS according the definition of the NCEP-ATPIII. Approximately 20% of adults had high blood pressure (hypertension), and 50% had a body mass index above 25 kg/m2.
  * The genetic and environmental determinants, through a multifaceted approach including familial segregation and candidate genes, the progression of cardiovascular risk and the incidence of cardiovascular diseases (vascular and coronary diseases, heart failure).

Methodology, Organization:

All Cohort members will be contacted to participate in this fourth visit. The data collected will be identical to those collected during the previous visits. However, they will be enriched with new clinical phenotyping conducted at the CIC (principal investigator Prof. Zannad): collection of blood and urine samples (DNA, RNA, lymphocytic extracts, plasma biobank, urology biobank), and morphological investigations (electrocardiogram, echocardiography, carotid echotracking, arterial stiffness, systolic pressure index, abdominal aortic ultrasound). Based on previous participation rates, the recruitment of 2,000 participants (500 families) is possible.

Expected Results:

This reconvening, for the follow-up at 17 years of the Stanislas Cohort, unique in its familial nature and having already contributed in a very significant manner in terms of knowledge generated, will enable in addition to the long-term continuation of its initial objectives (gene-environment interactions and cardiovascular diseases : Sophie Visvikis-Siest) to identify more specifically the natural history of the evolution of cardiovascular risk factors, including metabolic syndrome and its components as well as the incidence and transition mechanisms toward common cardiovascular diseases, notably vascular and coronary diseases and heart failure.

ANCILLARY STUDY

Detailed description of the ESCIF ancillary study - Dr. BONNEMAINS :

Objectives :

* to compare cardiac functional indices measured in MRI with the GRICS technique with equivalent indices measured with echocardiography.
* to assess inter-observer reproducibility of echography and MRI.

Organization :

76 subjects from the Stanislas cohort will be included prospectively in two groups according to the echocardiographic strains and tissue Doppler velocities acquired during echocardiography : 38 subjects with normal indices, and 38 with altered indices. Each subject will be proposed an MRI examination with the GRICS technique the same day to assess the same indices.

Study design = interventional: MRI. Prospective Number of groups: 2 Enrollment: 76 Last inclusion in the ESCIF study : 23/09/2014

SUBSTUDY : PHRC I 2013 - BioSe-PreIC - Dr HUTTIN : diagnostic performance of circulating biomarkers in early screening of heart failure Design : non interventionnal study

Main objective : Determine the contribution, in addition (ontop of ) of the subject's clinical characteristics, of circulating biomarkers assays (Gal-3, PIIINP, ST2) in a general population to screen early stages of heart failure (Stage B: asymptomatic patients with structural abnormalities) validated by trans-thoracic echocardiography (diastolic function and left ventricular mass)

Inclusion crieria :

Subjects participating to the 4th visit of the STANISLAS cohort

Subjets over 40 years old

Non-inclusion criteria :

Blood sample or echocardiography unavailable

Known cardiopathy

Modarate to severe sympptoms linked to heart failure

Présence of an abnormal diastolic function (E/Ea ratio above 8) and/or left ventricular hypertrophy (left ventricular mass above 125 g/m² for men and 110 g/m² for women).

ELIGIBILITY:
Inclusion Criteria:

* Patient having taken part in the STANISLAS troop,
* At least 18 years old,
* Written and signed enlightened assent,
* Ensured social

Exclusion Criteria:

* Patient unable to understand the informed consent,
* patient under legal protection

STANISLAS ancillary study:

Study population = subgroup of 76 subjects from the Stanislas cohort

Eligibility:

being member of the Stanislas cohort and participating to 4th visit Specific written and signed enlightened consent for the ESCIF study

Exclusion:

contraindications for MRI examination, possibility of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1705 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
investigating gene-gene and gene-environment interactions in the field of cardiovascular diseases | day 1
  study of inter-individual variability and familial segregation analysis of biological and morphological intermediate phenotypes of cardiovascular risk
ESCIF ancillary study : pair-wise comparison of functional indices measured in MRI and echocardiography | day 1

SECONDARY OUTCOMES:
ESCIF ancillary study : inter-observer reproducibility of each method (MRI and Echocardiography) | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Faiez ZANNAD, PU, PH, Principal Investigator — CHU Nancy, CIC-P, INSERM
Locations (2):
- France (2):
  - Centre d'Investigation Clinique -Plurithématique, Nancy
  - Centre d'Investigation Clinique- INNOVATIONS TECHNOLOGIQUES, Nancy

REFERENCES:
- [Derived] Lagrange J, Jahangiri M PhD, Baudry G, Mercier N, Monzo L, Lamiral Z, Duarte K, Ter Maaten JM, Zannad F, Voors AA, Girerd N. Association Between Endothelial Alterations, Cardiac Function, and Outcomes From Health to Heart Failure: Insight From the STANISLAS, MEDIA-DHF, and BIOSTAT-CHF Cohorts. J Am Heart Assoc. 2025 Jun 3;14(11):e040179. doi: 10.1161/JAHA.124.040179. Epub 2025 May 29. PMID 40439171
- [Derived] Lai TP, Verhulst S, Savage SA, Gadalla SM, Benetos A, Toupance S, Factor-Litvak P, Susser E, Aviv A. Buildup from birth onward of short telomeres in human hematopoietic cells. Aging Cell. 2023 Jun;22(6):e13844. doi: 10.1111/acel.13844. Epub 2023 Apr 28. PMID 37118904
- [Derived] Kobayashi M, Huttin O, Magnusson M, Ferreira JP, Bozec E, Huby AC, Preud'homme G, Duarte K, Lamiral Z, Dalleau K, Bresso E, Smail-Tabbone M, Devignes MD, Nilsson PM, Leosdottir M, Boivin JM, Zannad F, Rossignol P, Girerd N; STANISLAS Study Investigators. Machine Learning-Derived Echocardiographic Phenotypes Predict Heart Failure Incidence in Asymptomatic Individuals. JACC Cardiovasc Imaging. 2022 Feb;15(2):193-208. doi: 10.1016/j.jcmg.2021.07.004. Epub 2021 Sep 15. PMID 34538625
- [Derived] Monzo L, Ferreira JP, Lamiral Z, Bozec E, Boivin JM, Huttin O, Lopez-Sublet M, Girerd N, Zannad F, Rossignol P. Isolated diastolic hypertension and target organ damage: Findings from the STANISLAS cohort. Clin Cardiol. 2021 Nov;44(11):1516-1525. doi: 10.1002/clc.23713. Epub 2021 Sep 15. PMID 34523741
- [Derived] Wagner S, Lioret S, Girerd N, Duarte K, Lamiral Z, Bozec E, Van den Berghe L, Hoge A, Donneau AF, Boivin JM, Merckle L, Zannad F, Laville M, Rossignol P, Nazare JA. Association of Dietary Patterns Derived Using Reduced-Rank Regression With Subclinical Cardiovascular Damage According to Generation and Sex in the STANISLAS Cohort. J Am Heart Assoc. 2020 Apr 7;9(7):e013836. doi: 10.1161/JAHA.119.013836. Epub 2020 Mar 21. PMID 32200718
- [Derived] Benetos A, Verhulst S, Labat C, Lai TP, Girerd N, Toupance S, Zannad F, Rossignol P, Aviv A. Telomere length tracking in children and their parents: implications for adult onset diseases. FASEB J. 2019 Dec;33(12):14248-14253. doi: 10.1096/fj.201901275R. Epub 2019 Oct 25. PMID 31652401
- [Derived] Ferreira JP, Girerd N, Bozec E, Machu JL, Boivin JM, London GM, Zannad F, Rossignol P. Intima-Media Thickness Is Linearly and Continuously Associated With Systolic Blood Pressure in a Population-Based Cohort (STANISLAS Cohort Study). J Am Heart Assoc. 2016 Jun 16;5(6):e003529. doi: 10.1161/JAHA.116.003529. PMID 27312804